CLINICAL TRIAL: NCT03552406
Title: A Phase I, Open-label, Dose-finding Study to Assess the Safety, Tolerability and Pharmacokinetics of ISU104, a Human Monoclonal Antibody Targeting ErbB3 in Patients With Advanced Solid Tumors
Brief Title: Study of ISU104, Targeting ERBB3 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISU104-001
Record Dates: First submitted 2018-05-02; First posted 2018-06-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor
Keywords: Solid tumor; Breast cancer; Head & Neck cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms | interventions — Cetuximab; ErbB Receptors

STUDY DESIGN:
Intervention Model Description: A. Part 1: Dose escalation
  * Total 15 subjects: 3 subjects in each dose level
  * 1mg/kg/day, 3mg/kg/day, 5mg/kg/day, 10mg/kg/day, 20mg/kg/day
  B. Part 2: Dose expansion
  * Group 1 (Mono-therapy: 20 mg/kg/day, Q3W): 6 subjects
  * Group 2 (Combination therapy with cetuximab 400 mg/m2 followed by 250 mg/m2, Q1W): 12 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose-Escalation of ISU104 (Dose-Level 1) (Experimental): 1 mg/kg; Administered single-dose first week and observation for 4-weeks and then Administered once weekly in a 28-days Cycle
  Interventions: Biological: ISU104
- Dose-Escalation of ISU104 (Dose-Level 2) (Experimental): 3 mg/kg; Administered single-dose first week and observation for 4-weeks and then Administered once weekly in a 28-days Cycle
  Interventions: Biological: ISU104
- Dose-Escalation of ISU104 (Dose-Level 3) (Experimental): 5 mg/kg; Administered single-dose first week and observation for 4-weeks and then Administered once weekly in a 28-days Cycle
  Interventions: Biological: ISU104
- Dose-Escalation of ISU104 (Dose-Level 4) (Experimental): 10 mg/kg; Administered single-dose first week and observation for 4-weeks and then Administered once weekly in a 28-days Cycle
  Interventions: Biological: ISU104
- Dose-Escalation of ISU104 (Dose-Level 5) (Experimental): 20 mg/kg; Administered single-dose first week and observation for 4-weeks and then Administered once weekly in a 28-days Cycle
  Interventions: Biological: ISU104
- Dose-Expansion of ISU104 (Group 1: Monotherapy) (Experimental): ISU104 20 mg/kg to be administered every three weeks (Q3W) as monotherapy
  Interventions: Biological: ISU104
- Dose-Expansion of ISU104 (Group 2: Combination therapy) (Experimental): ISU104 20 mg/kg (or decreased dose) Q3W in combination with cetuximab* 250 mg/m2 QW (*Initial dose: 400 mg/m2)
  Interventions: Biological: ISU104; Drug: Cetuximab

INTERVENTIONS:
Biological: ISU104 — Intravenous Infusion for 1 hour.
  Other Names: A human monoclonal antibody targeting ErbB3
Drug: Cetuximab — Intravenous Infusion for 1 hour (2 hours at initial dose)
  Other Names: Erbitux; Epidermal Growth Factor Receptor (EGFR) inhibitor
  Arms: Dose-Expansion of ISU104 (Group 2: Combination therapy)

SUMMARY:
A phase I, open-label, dose-finding study to assess the safety, tolerability and pharmacokinetics of ISU104, a human monoclonal antibody targeting erbB3 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
[Part 1 Dose-escalation]

This study ams to evaluate the safety, tolerability, and pharmacokinetics of ISU104 in patients with advanced solid tumors.

Primary objective To determine recommended Phase II dose (RP2D) of ISU104 based on the results of its safety and tolerability in patients with advanced solid tumors.

Secondary objectives

1. To evaluate pharmacokinetics (PK) of ISU104 in patients with advanced solid tumors.
2. To evaluate efficacy of ISU104 in patients with advanced solid tumors.

Exploratory purpose To identify the expression of explorable multiple tumor biomarkers and to analyze the relationship between biomarkers and antitumor activity of ISU104.

[Part 2 dose-expansion] The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ISU104 in patients with recurrent/metastatic HNSCC (except for nasopharyngeal cancer), when administered intravenously ISU104 alone or ISU104 in combination with cetuximab.

Primary objective To determine RP2D of ISU104 based on results of its safety and tolerability in patients with recurrent/metastatic HNSCC (except for nasopharyngeal cancer), when administered intravenously ISU104 only or ISU104 in combination with cetuximab.

Secondary objectives

1. To evaluate the pharmacokinetics of ISU104 in patients with recurrent/metastatic HNSCC (except for nasopharyngeal cancer), when administered intravenously ISU104 only or ISU104 in combination with cetuximab.
2. To evaluate the efficacy of ISU104 in patients with recurrent/metastatic HNSCC (except for nasopharyngeal cancer), when administered intravenously ISU104 only or ISU104 in combination with cetuximab.

Exploratory purpose To explore a variety of detectable tumor biomarkers and evaluate the relationship between these biomarkers and antitumor activity of ISU104.

ELIGIBILITY:
Inclusion Criteria:

Common

1. Male or Female with ≥ 19 years of age
2. Histologically or Cytologically confirmed a diagnosis of an advanced solid tumor that was refractory to standard treatment or for which no standard therapy existed, or patients declined any treatment options
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Life Expectancy ≥ 12 weeks
5. Adequate Hematological, Renal and Hepatic function
6. According to Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1, the patient had at least one measurable lesion

Exclusion Criteria:

1. Severe hypersensitivity or a history of any hypersensitivity to the similar drug class of IP
2. Patients underwent the major surgery or procedure, or had the medical history (as blow):

   * Major surgery requiring systemic anesthesia or respiratory assist device within 4 weeks prior to baseline [2 weeks in case of video-assisted thoracoscopic surgery (VATS) or open-and-closed (ONC) surgery)]
   * Severe cardiovascular disease within 24 weeks prior to baseline
   * Severe cerebrovascular disease within 24 weeks prior to baseline
   * Pulmonary thromboembolism, deep vein thrombosis (DVT) or other clinically and significantly severe lung disease within 24 weeks prior to baseline
3. Patients had the following concurrent diseases at baseline:

   * Hematologic malignancies including lymphoma
   * Clinically significant symptom or uncontrolled central nervous system (CNS) or brain metastases
   * Pleural effusion and ascites drainage
   * Uncontrolled hypertension (SBP/DBP > 160/100 mmHg)
   * Active hepatitis B or C virus
   * Human immunodeficiency virus (HIV) that is positive
   * Thromboembolic disease or bleeding diatheses
   * Interstitial lung disease (ILD)
4. Left ventricular ejection fraction (LVEF) value, when measured by echocardiogram, multiple gated acquisition (MUGA) scan or a standard procedure in the institution within 4 weeks prior to the study entry
5. Patients with the following medication history:

   * anti-ErbB3 targeted therapies
   * small-molecule tyrosine kinase inhibitors within 2 weeks prior to baseline
   * any anti-cancer therapy, including chemotherapy, radiotherapy, biologic therapy, retinoid therapy, or therapeutic/palliative radiotherapy for the treatment of advanced solid tumors within 4 weeks prior to baseline
   * Granulocyte-Colony Stimulating Factor (G-CSF), packed red cell or platelet transfusion within 2 weeks prior to the first injection of IP to correct the abnormal values of absolute neutrophil count (ANC) or platelet count
6. Pregnant woman, breastfeeding woman, or women of childbearing age and men with partners of childbearing age, unless they are willing to follow abstinence or use effective forms of contraception* from the study entry until at least 16 weeks after the EOT visit
7. Subjects receiving any other investigational products or medical devices within 4 weeks prior to screening
8. Principal investigator's opinion

[Part 1 Dose-escalation cohort]

1. Patients with severe hypersensitivity or history of hypersensitivity to the similar drug class of the investigational product.
2. Patients receiving anti-cancer therapy, including chemotherapy, radiotherapy, biologic therapy, retinoid therapy, or therapeutic/palliative radiotherapy for treatment of advanced solid tumors within four weeks prior to baseline.

[Part 2 dose-expansion cohort]

1. Patients with history of allergy or hypersensitivity to the investigational product (ISU104 or cetuximab) or any excipients of the investigational product or its similar derivatives.
2. Patients with primary malignant neoplasm, including head and neck cancer as specified in inclusion criteria of Part 2 dose-expansion cohort. However, an exception may be allowed for the following:

   * For respective malignancy, treatment-naïve or disease-free patients for at least three years (however, patients undergoing radical resection on papillary thyroid carcinoma may be eligible for this clinical trial, even though three years have not passed).
   * Total dissection of skin basal cell carcinoma/squamous cell carcinoma or at least one year had passed since successful treatment of cervical intraepithelial neoplasia.
3. Patients receiving anti-cancer therapy, including chemotherapy, radiotherapy, biologic therapy, retinoid therapy, therapeutic/palliative radiotherapy, or hormone therapy for treatment of advanced solid tumors within four weeks prior to baseline.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose Dependent on Reports of Dose-limiting Toxicities | From date of first dose to 4 weeks after administration.
  Determination of MTD is dependent upon number of cohorts and patients required

SECONDARY OUTCOMES:
Toxicity Evaluation | through the study completion, an average of 1 year
  To determine the occurrence of Adverse Events (AEs)
Determine Immunogenicity of ISU104 | through the study completion, an average of 1 year
  To measure the level of Anti-Drug Antibody (ADA) and/or Neutralizing Antibody (NAb) of ISU104
Determine the Peak Plasma Concentration (Cmax) of ISU104 | up to 12 weeks
  To measure the Peak Plasma Concentration (Cmax) of ISU104
Determine the Area Under the Curve (AUC) of ISU104 | up to 12 weeks
  To measure the Area under the plasma concentration versus time curve (AUC) of ISU104
Explore Overall Response Rate (ORR) of ISU104 or ISU104+Cetuximab | up to progression, an average 6 months
  To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response (PR) is defined as >30% decrease in tumor burden from baseline and a Complete Response (CR) is defined as complete disappearance from tumor burden from baseline
Explore Disease Control Rate (DCR) of ISU104 or ISU104+Cetuximab | up to progression, an average 6 months
  To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response (PR) is defined as >30% decrease in tumor burden from baseline, a Complete Response (CR) is defined as complete disappearance from tumor burden from baseline, and Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for Partial Response nor sufficient increase to qualify for Partial Response (defined as >20% decrease in tumor burden from baseline)
Explore Progression-Free Survival (PFS) of ISU104 or ISU104+Cetuximab | up to progression, an average 6 months
  To measure the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

CONTACTS AND LOCATIONS:
Overall Officials: Jaehyeon Juhn, Ph.D, Study Director — ISU Abxis Co., Ltd.
Locations (5):
- South Korea (5):
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo S, Keam B, Shin SH, Chae YS, Kim TM, Park LC, Hong SB, Ahn MJ, Kim SB. A phase Ia/Ib study of novel anti-ErbB3 monoclonal antibody, barecetamab (ISU104) in refractory solid cancers and monotherapy or in combination with cetuximab in recurrent or metastatic head and neck cancer. Int J Cancer. 2023 Oct 15;153(8):1501-1511. doi: 10.1002/ijc.34622. Epub 2023 Jun 26. PMID 37357950